CLINICAL TRIAL: NCT04179279
Title: Comparative Analysis of a Non-contact Respiratory and Heart Rate Monitor Vs. a Conventional Clinically Validated Reference Monitor
Status: Completed | Type: Observational
Sponsor: ContinUse Biometrics Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CUBX-06
Record Dates: First submitted 2019-11-24; First posted 2019-11-27 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2019-11

CONDITIONS: Heart Rate; Respiratory Rate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pilot
  Interventions: Device: Gili Biosensor System (Gili Pro Biosensor)
- Pivotal
  Interventions: Device: Gili Biosensor System (Gili Pro Biosensor)

INTERVENTIONS:
Device: Gili Biosensor System (Gili Pro Biosensor) — Non-contact monitoring of heart and respiratory rates using an optical device

SUMMARY:
This is a prospective pivotal study in patients admitted/visiting the cardiology ward and/or outpatient clinics for various indications.

The study will be conducted in two stages. The first stage will comprise a pilot study with 10 subjects, which will be completed and analyzed prior to initiation of the second stage. The two studies are independent and are included in the same protocol for logistical reasons. The second stage of the study, which will include 120 subjects, is pivotal and intended to validate the Gili BioSensor System.

Testing procedure will include seating the subject in either a steady chair in front of a table, or in bed with the bedrest raised in front of a cardiac table (or similar). The subject will be seated for 5 minutes to reach a physiological steady state. During this time, the subject will be connected to the reference device according to the manufacturer's guidelines. The investigational device will be placed on a stable surface in front of the subject (table / cardiac table or similar) and will point to the left side of the subject's chest. Both the investigational and reference devices will be temporally synchronized to maintain coordinated recording. Following the 5-minute resting period, both investigational and reference devices will be activated for a comparative recording session to acquire at least 180 seconds (3 minutes) of evaluable data. Each 60-sec interval will be used separately for comparative analyses.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18, male or female
* Hemodynamically stable as assessed by the investigator
* Willing and able to sign informed consent

Exclusion Criteria:

* Inability to consent/comply with study protocol
* Presence of a condition that may interfere with the devices' performance (e.g. nausea, vomiting, persistent coughing, tremor, mouth breathing, etc.)
* Use of reflective garment, (e.g. sequin, silk, or similar), or highly textured garments (e.g. fur, thick lace, shaggy wool etc.).
* Parallel participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted/visiting the cardiology ward and/or outpatient clinics for various indications
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2019-10-06 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-01-27 (Actual)

PRIMARY OUTCOMES:
Heart rate | During the procedure
  Heart rate will be compared to a reference:
  * Accurate = 1 = device outcome is within ± 5 bpm or ± 10% bpm relative to reference, whichever is greater
  * Inaccurate = 0 = otherwise
Respiratory rate | During the procedure
  Respiratory rate will be compared to a reference:
  * Accurate = 1 = device outcome is within ± 2 breaths/min relative to reference
  * Inaccurate = 0 = otherwise

SECONDARY OUTCOMES:
Safety evaluation | During the procedure
  The Gili BioSensor System functions without physical contact with the inspected subject, and is compared in this study to a reference device routinely used as standard of care (SOC). Consequently, we do not expect any safety issues. At the same time, any adverse events (AE) observed during the procedure and/or during the study and/or follow-up period will be recorded in the CRF.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center (TASMC), Tel Aviv, Israel